CLINICAL TRIAL: NCT06302452
Title: ACTFAST: Urban and Rural Trauma Centers RE-AIM at Firearm Injury Prevention
Brief Title: Adult Trauma Centers RE-AIM at Gun Safety
Acronym: ACTFAST
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); Rhode Island Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: IRB00433605; R01MD019173 (NIH)
Record Dates: First submitted 2024-02-27; First posted 2024-03-08 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Firearm Injury; Safety Issues
MeSH Terms: interventions — Trauma Centers

STUDY DESIGN:
Intervention Model Description: The trial uses a unidirectional crossover stepped wedge design with a sequential roll-out of the intervention, ACTFAST, RE-AIM implementation framework, over several discrete time points or "steps." Each of the three trauma centers will be randomly assigned to one step that will determine when they crossover from control to implementation.
  Data are collected over multiple wedges, each 4-6 months in length. During the first wedge, none of the participating trauma centers will receive ACTFAST. During the second wedge, the first trauma center completes the Adoption and Implementation period. Over the third wedge, the first center shifts to the Maintenance period, the second trauma center enters the Adoption and Implementation period, and the remaining cohort stays in the control condition. This pattern continues until all trauma centers have progressed from control condition through the active implementation period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Intervention: Standard Care (No Intervention): All trauma patients will receive standard routine care which may include some screening and counseling on gun safety.
- ACTFAST Intervention (Experimental): During the implementation and maintenance periods, all trauma patients will receive study activities including firearm access screening, counseling on safe storage practices, and referral to safe storage and other community resources as appropriate.
  Interventions: Behavioral: Adopting Comprehensive Training for FireArm Safety in Trauma Centers

INTERVENTIONS:
Behavioral: Adopting Comprehensive Training for FireArm Safety in Trauma Centers — Firearm access screening, brief firearm safe storage intervention, and referral to community and preventive health resources
  Arms: ACTFAST Intervention

SUMMARY:
The goal of this interventional study is to evaluate the implementation and effectiveness of a comprehensive a universal firearm injury prevention program, ACTFAST (Adopting Comprehensive Training for FireArm Safety in Trauma centers), in level 1 trauma centers. The main aims of the study are:

1. (Primary Aim 1) Increase the adoption, implementation, and maintenance of a universal firearm injury prevention intervention at three participating trauma centers in the mid-Atlantic states;
2. (Primary Aim 2) Assess firearm injury prevention knowledge, attitudes, and safe storage practices among trauma patients treated within participating trauma centers.

ELIGIBILITY:
Electronic Medical Record (EMR) Participants:

Inclusion Criteria:

* trauma patients admitted to adult trauma inpatient services at participating institutions

Exclusion Criteria:

* none

Patient participants

Inclusion Criteria:

* at least 18 years of age;
* admitted to a participating trauma service for an injury;
* fluent in English or Spanish;
* able to provide informed consent.

Exclusion Criteria:

* prisoner or in police custody;
* admitted due to suicide attempt
* any acute conditions that would preclude provision of informed consent or assent (i.e., acute psychosis, altered mental status, cognitive impairment).

Staff participants

Inclusion Criteria:

* trauma service physician, physician assistant, nurse practitioner, nurse or social worker at participating pediatric trauma center

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1776 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of admitted injured patients receiving each element of the ACTFAST Program | 48 weeks
  ACTFAST components will be collected through retrospective data abstraction of each site's electronic medical record to determine if admitted injured patients received the Screening, Brief Intervention and Referral to Treatment (SBIRT) program components during the different phases of the study.
Percentage of admitted injured patients receiving elements of the ACTFAST Program | Admission, 2 weeks post discharge
  Among those eligible, compared to pre-implementation, there will be a difference in patients receiving each element of the ACTFAST program as measured by participant survey responses gathered during the participant's admission and 2-weeks post-discharge from survey data derived from multiple sources developed through the prior work of members of the study team.
Patient firearm safety attitudes and behaviors as assessed by survey | 48 weeks
  This outcome will be measured using the patient survey data adapted from prior work by the study team.

SECONDARY OUTCOMES:
Clinician firearm safety knowledge and confidence as assessed by survey | 48 weeks
  This outcome will be measured using clinician survey data derived from multiple sources developed through the prior work of members of the study team.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Hoops, MD, MPH, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No
At the conclusion of the study, deidentified data will be made publicly available. Due to the sensitive nature of the topics being discussed, individual participant data will not be made available to other researchers outside of the study team.